CLINICAL TRIAL: NCT00947960
Title: A Treatment Trial of Triheptanoin in Patients With Adult Polyglucosan Body Disease - A Randomized Controlled Study
Brief Title: Triheptanoin Treatment Trial for Patients With Adult Polyglucosan Body Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Baylor Research Institute (Other)
Collaborators: Ultragenyx Pharmaceutical Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 009-103
Record Dates: First submitted 2009-07-24; First posted 2009-07-28 (Estimated); Last update posted 2018-03-05 (Actual); Status verified 2018-03

CONDITIONS: Adult Polyglucosan Body Disease; Glycogen Brancher Enzyme Deficiency; Glycogen Storage Disease Type IV
Keywords: Adult Polyglucosan Body Disease (APBD); Glycogen Brancher Enzyme (GBE1) Deficiency
MeSH Terms: conditions — Polyglucosan Body Disease, Adult Form; Glycogen Storage Disease Type IV | interventions — triheptanoin; Plant Oils

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active/Placebo (Other): Subjects receive 1-2 grams/kilogram body weight triheptanoin divided into 4 equal doses taken with meals and snack for 6 months crossing over to receive placebo vegetable oil at the same dose and frequency for the next 6 months during the randomization phase.
  Interventions: Drug: Triheptanoin; Other: Vegetable Oil
- Placebo/Active (Other): Subjects receive 1-2 grams/kilogram body weight placebo vegetable oil divided into 4 equal doses taken with meals and snack for 6 months crossing over to receive triheptanoin at the same dose and frequency for the next 6 months during the randomization phase.
  Interventions: Drug: Triheptanoin; Other: Vegetable Oil

INTERVENTIONS:
Drug: Triheptanoin — 1-2 grams triheptanoin (drug)/kilogram body weight divided into 4 equal doses per day taken with meals and a snack for 6 months followed by 1-2 grams vegetable oil (placebo)/kilogram body weight divided into 4 equal doses per day taken with meals and a snack for 6 months.
Other: Vegetable Oil — 1-2 grams vegetable oil (placebo)/kilogram body weight divided into 4 equal doses per day taken with meals and a snack for 6 months followed by 1-2 g triheptanoin (drug)/kilogram body weight for 6 months.
  Other Names: Placebo

SUMMARY:
The purpose of the study is to determine if triheptanoin is an effective treatment for the symptoms of Adult Polyglucosan Body Disease.

DETAILED DESCRIPTION:
Adult polyglucosan disease is a progressive neurogenetic disorder characterized by neurogenic bladder, progressive difficulty with walking, and sensory abnormalities in the lower extremities which typically present in the 4th or 5th decade of life. The pathogenesis of the disease includes the accumulation of intracellular polyglucosan bodies (amylopectin-like polysaccharides) in the peripheral nerves as well as the central nervous system cells and is often associated with brancher enzyme deficiency which causes improper glycogen formation. It is hypothesized that decreased glycogen degradation leads to energy deficit in the nervous system cells. Therefore, anaplerotic therapy may supply needed substrate to the citric acid cycle to correct the energy deficit. This intervention may slow, halt or reverse the progression of the disease, for which there is no effective treatment. The trial involves 18 subjects ingesting a diet supplemented with triheptanoin, a 7 carbon triglyceride or a placebo of vegetable oil at a dose of 1-2 g/kg/24 hours in a randomized crossover controlled double blind study. The study lasts one year with patients receiving triheptanoin for 6 mo and the placebo oil for 6 mo. Safety monitoring includes urine organic acids and acyl carnitine profile.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of APBD by the presence of mutations of the GBE1 gene in both alleles or brancher enzyme deficiency
* Willing and able to travel to Dallas TX
* Able to tolerate dietary oil
* Able to provide informed consent

Exclusion Criteria:

* Intercurrent medical conditions that would confound the assessment of efficacy, such as HIV or diabetes
* Patients who are wheelchair bound
* Patients deemed unsuitable for the study by the investigator

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2009-06; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Distance traveled in six minute walk test | every three months

CONTACTS AND LOCATIONS:
Overall Officials: Raphael Schiffmann, M.D, M.H.Sc, Principal Investigator — Institute of Metabolic Disease
Locations (1):
- Department of Genetics, Groupe Hospitalier Pitié-Salpêtrière, Paris, France

REFERENCES:
- [Derived] Schiffmann R, Wallace ME, Rinaldi D, Ledoux I, Luton MP, Coleman S, Akman HO, Martin K, Hogrel JY, Blankenship D, Turner J, Mochel F. A double-blind, placebo-controlled trial of triheptanoin in adult polyglucosan body disease and open-label, long-term outcome. J Inherit Metab Dis. 2018 Sep;41(5):877-883. doi: 10.1007/s10545-017-0103-x. Epub 2017 Nov 6. PMID 29110179